CLINICAL TRIAL: NCT05827653
Title: A Double-blind, Randomized, Placebo-controlled, Multiple Ascending Dose (MAD) Study in Healthy Elderly Volunteers and Alzheimer's Disease (AD) Patients to Investigate the Safety and Tolerability, Pharmacokinetics (PK), and Pharmacodynamics (PD) Effects of Multiple Intravenous Infusions of NX210c
Brief Title: MAD Study of NX210c
Acronym: CHDR2235
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Axoltis Pharma (Industry)
Collaborators: Centre for Human Drug Research, Netherlands (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: AXO-CLI-210c-02; 2022-002868-76 (EudraCT Number)
Record Dates: First submitted 2022-12-08; First posted 2023-04-25 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Healthy Elderly

STUDY DESIGN:
Intervention Model Description: A double-blind, randomized, placebo-controlled, multiple ascending dose study to investigate the safety, tolerability, pharmacokinetics (PK) and pharmacodynamic effects of multiple intravenous infusions of NX210c. Two doses will be investigated.
  Subjects will participate for approx. 124 days; up to 84 days for screening, 26 days of treatment and 14 days Follow-up. As part of the screening process subjects will undergo MRI and Mini-Mental State Examination to establish normal cognitive capacity and exclude any major neurological condition. Blood for PK will be drawn as well as for biomarkers testing. A CNS battery of pharmacodynamic measures including EEG and MRI will be performed, as well as Lumbar punctures for cerebrospinal fluid drug concentration determination and biomarker testing.
  The study will be overseen by a safety review committee, sentinel dosing will be applied for each cohort. The rest of the cohort will be dosed if administration of NX210c is safe and well tolerated.
Who Masked: Participant, Investigator
Masking Description: Study is double-blind. Only personnel involved in randomization and creating reports to facilitate safe dose escalation, are planned to be unblinded during study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cohort 1_active (Experimental): Dose 1 NX210c
  Interventions: Drug: NX210c
- Cohort 1_placebo (Experimental): Placebo
  Interventions: Drug: Placebo
- Cohort 2_active (Experimental): Dose 2 (TBC) NX210c.
  Interventions: Drug: NX210c
- Cohort 2_placebo (Experimental): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NX210c — 3 times a week, for 28 days
  Arms: Cohort 1_active; Cohort 2_active
Drug: Placebo — 3 times a week, for 28 days
  Arms: Cohort 1_placebo; Cohort 2_placebo

SUMMARY:
This study will investigate the safety and tolerability of multiple intravenous infusions of NX210c with two ascending doses as well as NX210c pharmacokinetics (PK), and pharmacodynamics (PD) effects in healthy elderly subjects.

DETAILED DESCRIPTION:
The prevalence of neurocognitive disorders (NCD), including neurodegenerative diseases (NDDs) such as Alzheimer's disease (AD) is increasing. NDDs are most common and prevalent in elderly people worldwide and cause progressive neuronal dysfunction, toxicities, and death. These diseases lead to an irreversible weakening of all brain functions, including cognitive impairment. There is not one single cause of cognitive impairment but rather several factors that can contribute to trigger or accelerate cognitive decline.

Preclinical in vitro and in vivo data have shown that NX210c exhibits important properties, which may be suitable for the treatment of neurological disorders in humans. (i.e., neuroprotection, neuro-regeneration, synaptic transmission, positive effects on cognition, anti-neuroinflammatory action).

The First In Human Single Ascending Dose study has been completed. In that study, NX210 was administered and well tolerated. The current project is a multiple ascending dose (MAD) study and designed to investigate the safety, tolerability, PK and pharmacodynamics (PD) effects of multiple intravenous infusions of NX210c in two dose levels in healthy elderly subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male or female participants, as determined by the Investigator, based upon a medical evaluation including medical history, physical examination, neurological examination, MMSE, MRI, lab tests and ECG.
* Aged ≥ 55 years, inclusive at screening, and with a maximum weight of 110 kg.
* Body mass index (BMI) between 18 and 32 kg/m2, inclusive at screening.

Exclusion Criteria:

* Evidence of any history, or any active or chronic disease or condition that could interfere with, or for which the treatment of might interfere with, the conduct of the study, or that would pose an unacceptable risk to the subject in the opinion of the investigator
* History of any known neurologic disease, cognitive impairment, or diagnosed decline in cognitive function abnormal related to the age, or history of seizure, (significant) head trauma, loss of consciousness, or significant neuroimaging findings, including but not limited to any previously known or discovered abnormalities on screening brain MRI that evoke neurological diagnosis indicative of clinically significant abnormality

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2022-12-05 (Actual); Primary Completion 2023-04-29 (Actual); Study Completion 2023-10-02 (Actual)

PRIMARY OUTCOMES:
Severity and incidence of treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), suspected unexpected serious adverse reactions (SUSARs) | Up to 16 days after last dose
  Severity and incidence of treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), suspected unexpected serious adverse reactions (SUSARs)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Kremer, MD, PharmD, PhD, Principal Investigator — Centre For Human Drug Research
Locations (1):
- Centre for Human Drug Research, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No
Anonymized subject data to be shared based on reasonable request